CLINICAL TRIAL: NCT01401478
Title: Prospective, Open-label, Multicenter Effectiveness and Safety Observational Study of Zemplar in Patients With Stage 5 Chronic Kidney Disease and Hyperparathyroidism on Hemodialysis in the Russian Federation
Brief Title: Observational Program of Zemplar in Patients With End Stage Chronic Kidney Disease and Parathyroid Disorder on Hemodialysis in the Russian Federation
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Almedis (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-838
Record Dates: First submitted 2011-07-22; First posted 2011-07-25 (Estimated); Results first posted 2014-02-28 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Secondary Hyperparathyroidism
Keywords: Secondary Hyperparathyroidism; Chronic Renal Insufficiency
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stage 5 Chronic Kidney Disease: Planned for Zemplar administration due to secondary hyperparathyroidism

SUMMARY:
Eighty-six eligible participants with secondary hyperparathyroidism will be enrolled at thirteen sites in Russia. Planned therapy will be six months. Participants with Stage 5 Chronic Kidney Disease and with hyperparathyroidism on hemodialysis will be included into the study. Ability of Zemplar, (paricalcitol) to lower intact Parathyroid Hormone level will be assessed during the study.

DETAILED DESCRIPTION:
Eighty-six eligible participants with secondary hyperparathyroidism will be enrolled at thirteen sites in Russia. Study drug will be administered per local prescribing guidelines. Planned therapy is six months. Intact Parathyroid Hormone will be measured at the Screening visit. All participants who meet the inclusion criteria and fail to meet the exclusion criteria will be included in the study.

Adverse events will be monitored throughout the observation period (and up to 30 days after the last dose of Zemplar).

Ability of Zemplar to lower intact Parathyroid Hormone level will be assessed throughout the study. Proportion of participants with the level of intact Parathyroid Hormone 150 - 300 pg/mL was stated as primary endpoint. Calcium and Phosphorus elevation will be also measured throughout the study.

The selected population is representative in relation to those who will take Zemplar in routine practice. Participants with contraindications to Zemplar therapy (as per the local label) will not be included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. Chronic Kidney Disease stage 5 receiving hemodialysis
3. Authorization (Consent) for Use/Disclosure of Data signed by the patient
4. Planned prescription of Zemplar treatment due to fair clinical need and irrespectively of the participation in the current program according to the local label within 2 weeks after screening into the program
5. Screening intact Parathyroid Hormone level (measured not earlier than 1 month before first dose of Zemplar) between 300 and 900 pg/mL

Exclusion Criteria:

1. Contraindications to Zemplar as indicated in approved label, including but not limited to hypersensitivity, hypervitaminosis D (serum D3 level above 32 ng/mL), concomitant use of vitamin D or phosphates, lactation period, pregnancy
2. Any experimental drug within the period of 30 days before the inclusion into the program
3. Screening Ca x P > 65 mg˄2/dL˄2
4. Screening normalized serum total calcium > 10.2 mg/dL
5. Necessity for calcitonin maintenance oral or intravenous glucocorticoids, or other drugs that could have affected calcium or bone metabolism, other than females on stable estrogen and/or progestin therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis centers
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2011-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Strugovshchikov, MD, Study Director — AbbVie LLC
Locations (13):
- Russia (13):
  - Site Reference ID/Investigator# 57348, Al'met'yevsk
  - Site Reference ID/Investigator# 57347, Cheboksary
  - Site Reference ID/Investigator# 58347, Chelyabinsk
  - Site Reference ID/Investigator# 67404, Iakutsk
  - Site Reference ID/Investigator# 57344, Irkutsk
  - Site Reference ID/Investigator# 57346, Kazan'
  - Site Reference ID/Investigator# 58356, Moscow
  - Site Reference ID/Investigator# 58348, Moscow
  - Site Reference ID/Investigator# 57342, Novosibirsk
  - Site Reference ID/Investigator# 57364, Orenburg
  - Site Reference ID/Investigator# 57363, Saint Petersburg
  - Site Reference ID/Investigator# 69687, Samara
  - Site Reference ID/Investigator# 69688, Ulan-Ude

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stage 5 Chronic Kidney Disease
Started | 86
Completed | 55
Not Completed | 31
Not completed — Study drug not available | 6
Not completed — Adverse Event | 5
Not completed — Hyperphosphatemia | 5
Not completed — Lost to Follow-up | 5
Not completed — Kidney transplantation | 3
Not completed — Withdrawal by Subject | 3
Not completed — Blood samples not available | 1
Not completed — Hyperphosphatemia and adverse event | 1
Not completed — Low intact parathyroid hormone | 1
Not completed — Serious adverse event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Stage 5 Chronic Kidney Disease
Number analyzed (Participants) | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 86
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Participants] | 45.4 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 38
Region of Enrollment [Number; unit: participants]
  Russian Federation | 86

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Who Reached a Target Level of Intact Parathyroid Hormone (iPTH) (150-300 pg/mL) Post-baseline at Least Once During the Study
Description: The percentage of participants who had a post-baseline intact parathyroid hormone (iPTH) level in the range of 150 to 300 pg/mL at least once during the study was recorded.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stage 5 Chronic Kidney Disease
Number analyzed (Participants) | 86
Percentage of participants | 60.5 [49.3 to 70.8]

2. Secondary Outcome: Percentage of Participants Who Reached the Kidney Disease Improving Global Outcomes Target Level of Intact Parathyroid Hormone (iPTH) at Least Once During the Study
Description: The percentage of participants who reached the Kidney Disease Improving Global Outcomes target level of intact parathyroid hormone (iPTH) (defined as achievement of iPTH level 2 to 9 times the upper limit of normal) at least once during the study was recorded.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stage 5 Chronic Kidney Disease
Number analyzed (Participants) | 86
Percentage of participants
  Baseline | 57.0 [45.8 to 67.6]
  Post-baseline | 87.2 [78.3 to 93.4]

3. Secondary Outcome: Percentage of Participants Who Reached the Kidney Disease Improving Global Outcomes Target Level of Intact Parathyroid Hormone (iPTH) at Each Visit During the Study
Description: The percentage of participants who reached the Kidney Disease Improving Global Outcomes target level of intact parathyroid hormone (iPTH) (defined as the achievement of iPTH level 2 to 9 times the upper limit of normal) at each visit during the study was recorded.
Time Frame: 6 months
Population: The analysis for this outcome was based on the number of participants (55) who completed the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stage 5 Chronic Kidney Disease
Number analyzed (Participants) | 55
Percentage of participants
  Baseline | 49.1 [35.4 to 62.9]
  Visit 1 | 65.5 [51.4 to 77.8]
  Visit 2 | 45.5 [32.0 to 59.4]
  Visit 3 | 67.3 [53.3 to 79.3]
  Visit 4 | 40.0 [27.0 to 54.1]
  Visit 5 | 41.8 [28.7 to 55.9]
  Visit 6 | 49.1 [35.4 to 62.9]

4. Secondary Outcome: Percentage of Participants Who Developed Elevated Calcium (Ca) x Phosphate (P) (> 75 mg˄2/dL˄2) Levels at Least Once Post-baseline During the Study
Description: The percentage of participants who developed elevated calcium (Ca) x phosphate (P) (> 75 mg˄2/dL˄2) levels at least once post-baseline during the study was recorded.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stage 5 Chronic Kidney Disease
Number analyzed (Participants) | 86
Percentage of participants | 38.4 [28.1 to 49.5]

5. Secondary Outcome: Percentage of Participants Who Developed Elevated Calcium (Ca) x Phosphate (P) (> 75 mg˄2/dL˄2) Levels at Each Visit Post-baseline During the Study
Description: The percentage of participants who developed elevated calcium (Ca) x phosphate (P) (> 75 mg˄2/dL˄2) levels at each visit post-baseline during the study was recorded.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stage 5 Chronic Kidney Disease
Number analyzed (Participants) | 86
Percentage of participants
  Visit 1 | 12.8 [6.6 to 21.7]
  Visit 2 | 16.3 [9.2 to 25.8]
  Visit 3 | 16.3 [9.2 to 25.8]
  Visit 4 | 4.7 [1.3 to 11.5]
  Visit 5 | 7.0 [2.6 to 14.6]
  Visit 6 | 8.1 [3.3 to 16.1]

6. Secondary Outcome: Percentage of Participants Who Developed Elevated Normalized Total Calcium (> 11.2 mg/dL) at Least Once Post-baseline During the Study
Description: The percentage of participants who developed elevated normalized total calcium (> 11.2 mg/dL) at least once post-baseline during the study was recorded.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stage 5 Chronic Kidney Disease
Number analyzed (Participants) | 86
Percentage of participants | 10.5 [4.9 to 18.9]

7. Secondary Outcome: Percentage of Participants Who Developed Elevated Normalized Total Calcium (> 11.2 mg/dL) at Each Visit Post-baseline During the Study
Description: The percentage of participants who developed elevated normalized total calcium (> 11.2 mg/dL) at each visit post-baseline during the study was recorded.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stage 5 Chronic Kidney Disease
Number analyzed (Participants) | 86
Percentage of participants
  Visit 1 | 1.2 [0.0 to 6.3]
  Visit 2 | 2.3 [0.3 to 8.1]
  Visit 3 | 2.3 [0.3 to 8.1]
  Visit 4 | 4.7 [1.3 to 11.5]
  Visit 5 | 2.3 [0.3 to 8.1]
  Visit 6 | 0 [NA to NA] — Since there were no participants with elevated normalized total calcium at Visit 6, the 95% Confidence Interval is not applicable.

8. Secondary Outcome: Percentage of Participants Who Developed Hypercalcemia and Hyperphosphatemia Leading to Study Termination
Description: The percentage of participants who developed hypercalcemia (too much calcium in the blood) and hyperphosphatemia (too much phosphate in the blood) leading to study termination was recorded.
  Hypercalcemia was defined as calcium level greater than 11.2 mg/dL for more than 8 weeks, and hyperphosphatemia was defined as phosphate level greater than 6.5 mg/dL for more than 8 weeks.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stage 5 Chronic Kidney Disease
Number analyzed (Participants) | 86
Percentage of participants
  Hypercalcemia | 0 [NA to NA] — Since there were no participants with a calcium level greater than 11.2 mg/dL for more than 8 weeks during the study, the 95% Confidence Interval is not applicable.
  Hyperphosphatemia | 7.0 [2.6 to 14.6]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of study drug administration until 30 days or five half-lives following discontinuation of study drug. In addition, SAEs were collected from the time the participant signed the informed consent.
Arm/Group | Stage 5 Chronic Kidney Disease
Serious Adverse Events (participants affected / at risk) | 3/86
Other Adverse Events (participants affected / at risk) | 6/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 5 Chronic Kidney Disease (N=86)
Circulatory collapse (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Post procedural hematoma (Injury, poisoning and procedural complications) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 5 Chronic Kidney Disease (N=86)
Restless legs syndrome (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1
Pruritus generalized (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.